CLINICAL TRIAL: NCT05030935
Title: Assessing the Feasibility of a Novel Preventive Mobile Health App Among Informal Caregivers of Outpatients at Risk of Developing Pressure Ulcers: A Quasi-Experimental Study
Brief Title: Assessing the Feasibility of a Prevention m-Health App Intervention for Informal Caregivers of Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nicosia (Other)
Responsible Party: Principal Investigator, Giannis Polychronis, Doctoral Candidate, University of Nicosia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ΕΕΒΚ/ΕΠ/2021/55
Record Dates: First submitted 2021-08-22; First posted 2021-09-01 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Telemedicine; Caregivers; Pressure Ulcer
Keywords: Pressure Ulcer Prevention, mHealth, quasi-experimental
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will be able to use the mHealth App.
  Interventions: Device: mHealth App
- Control group (No Intervention): The Instructions Manual consists of a hard copy of the mHealth App bibliographical content. In addition, a calendar that can be used as a reminder for patient position switching is present and a hard copy explanation of the scale which can be used by the caregiver and through handwriting, determine the need for support surfaces.

INTERVENTIONS:
Device: mHealth App — In short, mHA contains three main functions for the user: a) a reminder for switching the patient position, b) training for preventive care habits and c) the possibility for patient evaluation in order to determine the need for the use of support surfaces.
  Arms: Intervention Group

SUMMARY:
The present quasi-experimental study aims to compare the level of preventive behaviours amongst caregivers who will be instructed to operating one mHealth App or given a relevant instruction manual. To achieve this, a comparison between the behavior of caregivers before and after the intervention and a comparison between the two groups (intervention group with the control group) will be performed. Specifically, data within the two groups will be collected via an online questionnaire consisting of three parts: prior to the intervention (baseline), two (2) and four (4) months after the intervention. The self-administered questionnaire consists of fifty-two (52) questions and uses three valid and reliable scales with a part that was developed via a bibliography research and consultations from experienced specialists. The questionnaire scales have been translated from the English language to Greek.

ELIGIBILITY:
Inclusion Criteria:

* The main adult caregiver is able to provide care / support to a bedridden patient.
* Willingness to participate in the study.
* Basic knowledge of the Greek language such that the user can understand the intervention and be able to complete the self-administered questionnaire.
* Possession of a mobile Android or iOS device.
* The patient is bedridden for no longer than four (4) months.
* During the assessment for predicting the risk of patient PUs development, the score according to the BRADEN scale must be between medium to severe risk (≤ 18).

Exclusion Criteria:

* The user does not have basic knowledge of the Greek language such that he/she is not able to understand the intervention or complete the self-administered questionnaire.
* Possession of a different mobile device other than Android and iOS or no possession of a mobile device.
* The patient is bedridden for four (4) months or longer.
* A mild risk score using the BRADEN scale (15-18).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
FCAT: The Family Caregiver Activation in Transitions® | 4 months
  Change from baseline score (t1) of FCAT scale at 2 months measured (t2) and 4 months measured (t3) for both groups.
Pressure Ulcers Prevention Behaviors (PUPB) | 4 months
  Change from baseline (t1) of PUPB score at 2 months measured (t2) and 4 months measured (t3) for both groups.

SECONDARY OUTCOMES:
TAM: Technology Acceptance Model | 4 months
  Change from baseline score (t1) of TAM scale at 2 months measured (t2) and 4 months measured (t3) for intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Roupa, PhD, Study Director — University of Nicosia
Locations (1):
- University of Nicosia, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polychronis, G. et al. (2022) "A Pressure Ulcer Prevention mHealth App for Informal Caregivers of Bedridden Outpatients: Validation," Cyprus Nursing Chronicles, 22(2), pp. 9-18.